CLINICAL TRIAL: NCT02680613
Title: Pilot Study of a Mobile Health Approach to Reduce Barriers to Cervical Cancer Screening in Tanzania
Acronym: KCCPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Terry Fox Foundation (Other)
Responsible Party: Principal Investigator, Dr. Karen Yeates, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Q-6015511
Record Dates: First submitted 2016-02-09; First posted 2016-02-11 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Cervical Cancer
Keywords: Behaviour Change; Secondary Prevention; mHealth
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The participants were not aware of which group they were randomized to. The care provider providing the screening service was not aware of the group of the participant.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Motivational SMS (Experimental): This arm will receive 15 motivational SMS about cervical cancer and screening.
  Interventions: Behavioral: Motivational SMS
- Travel Voucher (Experimental): This arm will receive a voucher covering return transport from the screening clinic. This arm will also receive identical 15 motivational SMS about cervical cancer and screening as the Motivational SMS arm.
  Interventions: Behavioral: Motivational SMS; Behavioral: Travel Voucher
- Control (No Intervention): This arm will receive standard sensitization during study period (church announcements, screening promotion by key community leaders and posters in community, as well as sensitization by the research assistants conducting the door-to-door household recruitment) during the study and follow-up period. They will also receive one SMS message with the location of screening services during the study period. At the conclusion of the study, participants in the arm will receive identical motivational SMS as the other two arms.

INTERVENTIONS:
Behavioral: Motivational SMS — Behaviour change messages delivered via SMS developed with the theoretical guidance of the Health Belief Model.
  Arms: Motivational SMS; Travel Voucher
Behavioral: Travel Voucher — A code for return public transportation to closest cervical cancer screening clinic included in the research.
  Arms: Travel Voucher

SUMMARY:
The purpose of this study is to determine whether motivational text messages and/or travel vouchers are effective in increasing cervical cancer screening rates in urban and rural regions of Northern Tanzania.

DETAILED DESCRIPTION:
Introduction:

Cervical cancer is the leading cause of cancer-related deaths in Tanzania. The age-adjusted incidence rate is estimated to be 54 cases per 100,000 (IARC, 2012) and 80% of Tanzanian women affected by cervical cancer will die due to advanced stage at diagnosis (Kahesa, et al., 2012). Visual Inspection of the cervix under Acetic Acid (VIA) is an effective alternative to the Pap smear, unavailable in most low-resource countries due to weak health systems (Palanuwong, 2007). Nurses typically receive 6 days of training before returning to their communities to provide VIA; however, they often face a total lack of oversight to ensure they are providing quality screening and cryotherapy. This lack of quality control has prevented a decline in cervical cancer morbidity and mortality despite significant investment and implementation of VIA programs.

The Kilimanjaro Cervical Cancer Screening Project (KCCP) is a pilot study of 1000 women that developed and tested a cervicography (taking a digital photo of the cervix) training method using a smartphone camera in the hands of nurses performing cervical cancer screening and receiving 'real time' mentorship through a closed user group of image transfer and guidance by cervicographers located elsewhere in Tanzania. A pilot study completed in February 2015 showed that this method provides safe and high quality screening and the method is moving to implementation and scale up within multiple VIA programs in late 2015 (Yeates et al., Manuscript in preparation). The KCCP continues to screen patients and this provides a significant opportunity to perform further research that will inform the scale-up program.

Measures to encourage increased uptake of cervical cancer screening in the region, and in many low-resource contexts are drastically needed to reduce the burden of cervical cancer in these contexts. The prevalence of screening in the Kilimanjaro is 6%(Cunningham et al, 2015), which is close to the WHO figure of 5% of women in developing countries having been screened in the last five years (World Health Organization, 1986). The largest perceived barriers to cervical cancer screening in the Kilimanjaro region were found to be a lack of knowledge that screening services were available and women anticipated that they would not be able to afford the costs associated with screening, including travel (Cunningham et al, 2015).

Objectives:

A) To determine attitudes, barriers and enablers towards smartphone cervicography to ensure an accessible, culturally relevant smartphone cervicography screening program

B) To evaluate the impact of a voucher for return transportation towards increasing cervical cancer screening attendance

C) To evaluate the impact of motivational text messages towards increasing cervical cancer screening attendance

Methodology:

This study will comprise of a descriptive cross-sectional survey and a randomized controlled trial (RCT). Household surveys, capturing baseline characteristics, using stratified systematic random sampling in urban and rural areas will be used to recruit participants for the RCT. Cross-sectional survey participants will be recruited opportunistically at screening clinics associated with the study.

RCT participants will be randomized into one of three arms. The first arm will be a control group and will not receive any correspondence. The second arm will receive a series of motivational text messages, including screening dates and locations. The third group will receive a travel voucher code via SMS and motivational text messages with the same content as the second group.

A post-screening survey will be conducted following cervical cancer screening at clinics participating in the study to evaluate screening attendance and attitudes towards smartphone digital cervicography.

ELIGIBILITY:
Inclusion Criteria:

* Own a mobile phone or have access to husband's/friend's mobile phone who is not eligible to participate in the research

Exclusion Criteria:

* Previous history of cervical cancer or hysterectomy
* Having been screened for cervical cancer in the past year

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 851 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05-12 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Attendance at Cervical Cancer Screening at clinics included in Trial | within 60 days from recruitment into study
  The primary outcome is binary. It is whether or not participants attend cervical cancer screening at the clinics included in the randomized controlled trial.

SECONDARY OUTCOMES:
Satisfaction with Smartphone Enhanced Digital Cervicography | Completed if a client attended cervical cancer screening within the follow-up period (within 2 months of randomization)
  The secondary outcome is measured by two survey questions that were part of a exit-survey completed women following cervical cancer screening using the Smartphone Enhanced Visual Inspection with Acetic Acid (SEVIA) used at the two screening clinics included in our trial. The client is considered satisfied if they answer "Yes" to the question "Did you feel comfortable with having a photo of your cervix taken at screening?" and "Definitely Agree" or "Agree" to the question "Did reviewing the picture of your cervix at screening and using it to discuss your risks for cancer increase your knowledge of your risk of cancer?". Otherwise the client is considered dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Yeates, MD, Principal Investigator — Queen's University
Locations (1):
- Pamoja Tunaweza Women's Center, Moshi, Kilimanjaro, Tanzania

REFERENCES:
- [Background] Cunningham MS, Skrastins E, Fitzpatrick R, Jindal P, Oneko O, Yeates K, Booth CM, Carpenter J, Aronson KJ. Cervical cancer screening and HPV vaccine acceptability among rural and urban women in Kilimanjaro Region, Tanzania. BMJ Open. 2015 Mar 10;5(3):e005828. doi: 10.1136/bmjopen-2014-005828. PMID 25757944
- [Background] Kahesa C, Kjaer S, Mwaiselage J, Ngoma T, Tersbol B, Dartell M, Rasch V. Determinants of acceptance of cervical cancer screening in Dar es Salaam, Tanzania. BMC Public Health. 2012 Dec 19;12:1093. doi: 10.1186/1471-2458-12-1093. PMID 23253445
- [Background] World Health Organization, International Agency for Research on Cancer (IARC) (2012). WHO 2012 estimated cancer incidence, mortality and prevalence in 2012 Available at: http://globocan.iarc.fr/Pages/fact_sheets_population.aspx Accessed February 25, 2015
- [Background] Palanuwong B. Alternative cervical cancer prevention in low-resource settings: Experiences of visual inspection by acetic acid with single-visit approach in the first five provinces of Thailand. Aust N Z J Obstet Gynaecol. 2007 Feb;47(1):54-60. doi: 10.1111/j.1479-828X.2006.00680.x. PMID 17261102
- [Background] Yeates KE, Sleeth J, Hopman W, Ginsburg O, Heus K, Andrews L, Giattas MR, Yuma S, Macheku G, Msuya A, Oneko O. Evaluation of a Smartphone-Based Training Strategy Among Health Care Workers Screening for Cervical Cancer in Northern Tanzania: The Kilimanjaro Method. J Glob Oncol. 2016 May 4;2(6):356-364. doi: 10.1200/JGO.2015.001768. eCollection 2016 Dec. PMID 28717721
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] Erwin E, Aronson KJ, Day A, Ginsburg O, Macheku G, Feksi A, Oneko O, Sleeth J, Magoma B, West N, Marandu PD, Yeates K. SMS behaviour change communication and eVoucher interventions to increase uptake of cervical cancer screening in the Kilimanjaro and Arusha regions of Tanzania: a randomised, double-blind, controlled trial of effectiveness. BMJ Innov. 2019 Jan;5(1):28-34. doi: 10.1136/bmjinnov-2018-000276. Epub 2019 Feb 22. PMID 31645991